CLINICAL TRIAL: NCT00918853
Title: Prospective Evaluation of the Resection Margins and the Ganglionic Status Using a Quality Standard Resection for Adenocarcinoma of the Head of the Pancreas.
Acronym: MRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRP/IPC 2007-005; ID-RCB 2007-A01326-47
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Pancreas; Adenocarcinoma
Keywords: pancreas; adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- resection for adenocarcinoma (Experimental): quality standard resection for adenocarcinoma of the head of the pancreas
  Interventions: Procedure: resection of adenocarcinoma of the head of the pancreas

INTERVENTIONS:
Procedure: resection of adenocarcinoma of the head of the pancreas — quality standard for the resection of adenocarcinoma of the head of the pancreas

SUMMARY:
This multicentric prospective study evaluates the role of the margins resection and the ganglionic status when using a quality standard for the resection of adenocarcinoma of the head of the pancreas.

DETAILED DESCRIPTION:
Primary objective:

* Evaluation of the prognosis role of the invasion of the margins on the overall survival after a standard resection of adenocarcinoma of the head of the pancreas.

Secondary objectives:

* Evaluation of the prognosis role of the invasion:

  * Of margins on the overall survival.
  * Of each margins (distal pancreatic margin, gastric, posterior, retro-venous, retro-arterial) on the overall survival.
  * Of the ganglionic group of the superior mesenteric artery and the other nodes.

ELIGIBILITY:
Inclusion Criteria:

* A head of the pancreas tumor compatible with adenocarcinoma diagnosis
* tumor apparently removable
* patient aged from 18 to older
* signed consent

Non inclusion criteria:

* pregnancy, breast feeding
* patient in an urgency situation or patient with legal protection

Exclusion Criteria after surgery:

* tumor other than adenocarcinoma of the head of the pancreas.
* analysis of the margins not done with the defined criteria
* nonadhesion to the surgical protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Prognostic value of the invasion of the margins measured in millimetres on the overall survival | 4 years

SECONDARY OUTCOMES:
Relapse free survival: time between surgery and relapse or a right censure. The relapse is determined by clinical examination, biologic examination and imaging, which reveals metastasis or an isolated local relapse | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean Robert DELPERO, PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (20):
- France (20):
  - Chu D'Angers, Angers
  - Chu de Bordeaux, Bordeaux
  - Hopital Ambroise Pare, Boulogne
  - Chu de Clermont-Ferrand, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Hopital Henri Mondor, Créteil
  - Hopital de L'Antiquaille, Lyon
  - Hopital de La Croix-Rousse, Lyon
  - Hospices Civils de Lyon, Lyon
  - Chu La Conception, Marseille
  - Institut Paoli-Calmettes, Marseille
  - Centre Val D'Aurelle Paul Lamarque, Montpellier
  - Hotel Dieu, Nantes
  - Hopital Cochin, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Tenon, Paris
  - Hopitial Saint Antoine, Paris
  - Hopital Pontchaillou, Rennes
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Chu Purpan, Toulouse

REFERENCES:
- [Derived] Delpero JR, Jeune F, Bachellier P, Regenet N, Le Treut YP, Paye F, Carrere N, Sauvanet A, Adham M, Autret A, Poizat F, Turrini O, Boher JM. Prognostic Value of Resection Margin Involvement After Pancreaticoduodenectomy for Ductal Adenocarcinoma: Updates From a French Prospective Multicenter Study. Ann Surg. 2017 Nov;266(5):787-796. doi: 10.1097/SLA.0000000000002432. PMID 28953554
- [Derived] Delpero JR, Bachellier P, Regenet N, Le Treut YP, Paye F, Carrere N, Sauvanet A, Autret A, Turrini O, Monges-Ranchin G, Boher JM. Pancreaticoduodenectomy for pancreatic ductal adenocarcinoma: a French multicentre prospective evaluation of resection margins in 150 evaluable specimens. HPB (Oxford). 2014 Jan;16(1):20-33. doi: 10.1111/hpb.12061. Epub 2013 Mar 7. PMID 23464850
- See also: OFFICIAL WEB SITE OF THE SPONSOR — http://www.institutpaolicalmettes.fr/